CLINICAL TRIAL: NCT03721120
Title: A Randomized Phase III Clinical Trial to Evaluate the Feasibility and Clinical Relevance of Liquid Biopsy in Patients With Suspicious Metastatic Lung Cancer
Brief Title: Evaluation of the Feasibility and Clinical Relevance of Liquid Biopsy in Patients With Suspicious Metastatic Lung Cancer
Acronym: LIBELULE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ET18-086 LIBELULE
Record Dates: First submitted 2018-10-17; First posted 2018-10-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liquid biopsy (Experimental): Liquid biopsy will be performed at the first visit using InVisionFirst®. Treatment will be determined by (i) genomic characterization in plasma for patients with druggable alteration in first-line, (ii) after pathology results (including assessment of PD-L1 level of expression by immunohistochemistry) for patients with an informative molecular characterization on plasma and no druggable alteration in first-line and (iii) after pathology results and tissue molecular characterization for the remaining patients.
  Interventions: Diagnostic Test: InvisionFirst® molecular panel
- Cytological or histological sampling (No Intervention): During the first visit, cytological or histological sampling will be planned and treatment will be initiated according to European Society of Medical Oncology (ESMO) recommendations; in case of a tissue sample inadequate for genomic characterization, physicians may resort to liquid biopsy according to their usual practice and available technology.

INTERVENTIONS:
Diagnostic Test: InvisionFirst® molecular panel — During the first visit, liquid biopsy will be performed using the InVisionFirst® panel. Cytological or histological sampling will be planned. According to InVisionFirst® results, treatment will be initiated:
  * regardless of cytological/histological and tissue molecular analysis in case of EGFR, BRAF V600E-mutation, ALK- or ROS1-rearrangement identified on InvisionFirst® panel.
  * regardless of molecular characterization performed on tissue sample in case of ERBB2-, BRAF non V600E-, c-MET-, KRAS-,LKB1-, NTRK and/or RET mutation on InVisionFirst® panel. Treatment will be based on pathology results and if appropriate on PD-L1 level of expression.
  * for patients with none of the previous alterations, treatment will be initiated after obtaining pathology results and genomic characterization from the tumor tissue analysis.
  Arms: Liquid biopsy

SUMMARY:
Lung cancer is diagnosed at metastatic stage in 60% of the cases. For these patients, first-line treatment is based on histology and molecular characterization of non-squamous non-small cell lung cancer (NSCLC). Thus, quality and quantity of tumor tissue are crucial to determine the appropriate treatment (targeted therapies, chemotherapy and immunotherapy).

However, in routine practice, tissue quality and quantity can be limited (25%), resulting in the need for tumor rebiopsy for molecular analysis. Therefore, lung cancer patients often experience substantial delays before treatment initiation that may be associated with worse patient experience of subsequent cancer care and poorer clinical outcomes.

"Liquid biopsies" (LB) are used to detect genomic alterations in cell-free circulating DNA (cfDNA). Since very recently, they are routinely used in reference centers for the detection of EGFR-mutations when tissue is not sufficient for molecular characterization. Importantly, the feasibility and clinical relevance of systematic liquid biopsies in routine practice has never been evaluated in patients with suspicious advanced lung cancer.

Investigators hypothesize that using systematic LB in patients with clinical suspicion of metastatic lung cancer may reduce time-to-treatment initiation and avoid tissue rebiopsy.

Investigators performed a retrospective study including 250 NSCLC patients treated in a tertiary Cancer Center and in the University Hospital of Lyon, France. The mean time-to-appropriate frontline treatment initiation (TTI) was 42+/-22.5 days. With the use of LB at the time of first consultation, the investigators believe it is possible to reduce the mean TTI down to 33 days (21% reduction in TTI) in the overall population with suspicious metastatic lung cancer, including a 50% and 40% reduction in TTI for EGFR/ALK/ROS1/BRAF V600E subgroups and KRAS/LKB1/ERBB2/c-MET/BRAF non V600E subgroups, respectively.

Investigators therefore designed a "real-life" randomized study to evaluate the feasibility and clinical relevance of LB to decrease the TTI, which may in turn improve patients' outcome. Genomic analyses of circulating cfDNA will be performed using a robust and highly sensitive technology (InVision®), that profiles the presence of genomic aberrations in a panel of 35 genes including mutations, insertion/deletions and rearrangements, including all actionable alterations required to initiate the appropriate first-line therapy (EGFR-, ALK-, ROS1 and BRAF V600E).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with clinico-radiological suspicious presentation of stage IV lung cancer;
* No prior chemotherapy for locally advanced or metastatic NSCLC;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 (Appendix 2);
* Life expectancy > 12 weeks;
* No contraindication to systemic lung cancer treatment;
* Covered by a medical insurance;
* Signed informed consent prior to any study-specific procedure;
* No prior biopsy or cytology for lung cancer diagnosis.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Patient concurrently using other approved or investigational antineoplastic agents;
* Major concurrent disease affecting cardiovascular system, liver, kidneys, hematopoietic system or else considered as clinically important by the investigator and that could be incompatible with patient's participation in this trial or would likely interfere with study procedures or results;
* Prior history of malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease for at least 3 years;
* Patient requiring tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Time-to-appropriate Treatment Initiation (TTI) | From date of randomisation to start date of appropriate treatment , assessed up to 12 months
  It is defined as the time between the date of randomization and the date of appropriate-treatment initiation (whatever the start date occurs before or after the biopsy results). As all the patients will receive an appropriate-treatment, no censored data are expected, thus the TTI will be analyzed as a continuous outcome. Appropriate treatment is defined as follow:
  * Based on contributive results on tissue OR liquid biopsy:
    * EGFR- or BRAF V600E-mutations, ALK- or ROS1- rearrangements: specific targeted therapies
    * None of the four previous alterations: investigator's choice (chemotherapy and/or immunotherapy or targeted therapies based on pathology results, PD-L1 expression and access to therapies in the context of Temporary Used Authorization or clinical trials)
  * In case of non-contributive results on tissue AND liquid biopsy: any treatment initiated by investigator (chemotherapy or immunotherapy based on pathology results and PD-L1 level of expression).

SECONDARY OUTCOMES:
Rate of treatment initiated before molecular results | From date of randomisation to 12 months
  Defined as the proportion of patients with a treatment initiated without any available molecular results (tissue and liquid biopsy)
Time to availability of informative molecular pathology results | From date of randomisation to date of molecular results, assessed up to 12 months
  Defined as the time from randomization to date of availability of informative molecular pathology results (positive or negative).
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
  Defined as the time from randomization to the date of the first documented clinical or radiological progression (as per RECIST version 1.1.) or death due to any cause.Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment.
Incidence of diagnostic test-emergent adverse events | From date of randomization to follow-up visit month 12 or death due to any cause, whichever came first, assessed up to 30 months
  Safety assessed according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version5
The impact of cancer on the patient's quality of life using the European Organisation for Research and Treatment of Cancer (EORTC) quality-of-life core questionnaire (QLQ-C30) | At baseline, at Day 21 post-baseline, at the time of treatment initiation (within 6 weeks after baseline), at 8 weeks post treatment initiation and every 3 months post initiation of treatment until 12 months
  64 questions related to cancer impact on health and daily activities composed this questionnaire. Each item has to be graded from 1 to 4 (1 = not at all, 4= very much). More the score is high, worst the quality of life is.
Evaluation of lung cancer symptoms impact on health and daily activities using the Lung Cancer Symptoms Scale (LCSS) questionnaire | At baseline, at Day 21 post-baseline, at the time of treatment initiation (within 6 weeks after baseline), at 8 weeks post treatment initiation and every 3 months post initiation of treatment until 12 months
  10 questions related to lung cancer symptoms impact on health and daily activities composed this questionnaire. Each item has to be graded from 1 to 10. More the score is high, worst the quality of life is.
Evaluation of anxiety and depression level using Hospital Anxiety and Depression (HAD)Scale | At baseline, at Day 21 post-baseline, at the time of treatment initiation (within 6 weeks after baseline), and at 8 weeks post treatment initiation
  6 questions related to anxiety and 6 questions related to depression composed this questionnaire. Each item has to be graded from 0 to 3. More the score of anxiety or depression is high, worst the quality of life is.
Concordance between molecular status on tissue and liquid biopsies in the experimental arm | From date of randomization to follow-up visit month 12 or death due to any cause, whichever came first, assessed up to 30 months
  Evaluated by the proportion of discordances (error rates) between tissue and liquid biopsies for the mutational status.
Biopsy avoidance rate in the experimental arm | From date of randomization to follow-up visit month 12 or death due to any cause, whichever came first, assessed up to 30 months
  Be defined as the proportion of patients with an initial non-informative tissue biopsy and an informative liquid biopsy allowing appropriate treatment initiation without need for tissue rebiopsy.
The cost analysis | From date of randomization to follow-up visit month 12 or death due to any cause, whichever came first, assessed up to 30 months
  All costs items related to the stratégies and supported by the payers will be collected prospectively for each patient. Mean total costs will be calculated for the 2 stratégies and be compared between the arms.
The effectiveness analysis using the EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L) | At baseline, at Day 21 post-baseline, at the time of treatment initiation (within 6 weeks after baseline), at 8 weeks post treatment initiation and every 3 months post initiation of treatment until 12 months
  Preferences will be measured using EuroQoL 5 Dimensions 5 Levels questionnaire. Five attributes will therefore be investigated: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each attributes having five levels (from "able to […]"/"no pain/discomfort/anxiety/depression" to "unable to […]"/ "extremely pain/discomfort/anxiety/depression"). More the patient is unable to doing daily activities and painful/anxious, worst the quality-adjusted life-year (QALYs) is.
QALYS comparaison between 2 arms | At baseline, at Day 21 post-baseline, at the time of treatment initiation (within 6 weeks after baseline), at 8 weeks post treatment initiation and every 3 months post initiation of treatment until 12 months
  Mean QALYs (based on EQ-5D-5L score) will be calculated for each arm and will be compared between the 2 arms.
The budget impact analysis in experimental arm | From date of randomization to follow-up visit month 12 or death due to any cause, whichever came first, assessed up to 30 months
  The Liquid biopsy using the InVisionFirst® cost, the evolution of market shares, the data pertaining to the target population, and the costs involved with treating the pathologies will be analysed to to estimate the budget impact on the French National Health Insurance of the generalization of innovative Liquid biopsy using the InVisionFirst® panel strategy.
Exploratory objectives : Whole-exome sequencing | At baseline, at the time of treatment initiation (within 6 weeks after baseline), at 8 weeks after the treatment initiation, and at the progression if occured within 12 month post-baseline.
  Additional mandatory 10 ml DNA STRECK tubes will be collected for patients signing study consent.
Exploratory objectives : miRNA profiling | At baseline, at the time of treatment initiation (within 6 weeks after baseline), at 8 weeks after the treatment initiation, and at the progression if occured within 12 month post-baseline.
  Additional mandatory 10 ml RNA STRECK tubes will be collected for patients signing study consent.

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Centre Hospitalier de Bayeux, Bayeux
  - Hopital Louis Pradel, Bron
  - Centre François Baclesse, Caen
  - Centre Maurice Tubiana, Caen
  - Infirmerie Protestante, Caluire-et-Cuire
  - Centre Hospitalier Public du Cotentin, Cherbourg
  - CH Les Oudairies, La Roche-sur-Yon
  - Hôpital Privé Jean Mermoz, Lyon
  - Centre Leon Berard, Lyon
  - Groupe Hospitalier de la région de Mulhouse et Sud-Alsace, Mulhouse
  - Centre Hospitalier Annecy Genevois, Pringy
  - CHRU Saint-Etienne, Saint-Etienne
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Hôpital Nord-Ouest, Villefranche-sur-Saône
  - Médiôle Lyon-Villeurbanne, Villeurbanne